CLINICAL TRIAL: NCT04622254
Title: A Prospective, Randomized, Double-blind, Placebo-controlled, Multicenter Study With an Open-label Extension Period to Investigate the Efficacy and Safety of NT 201 in the Simultaneous Treatment of Upper Facial Lines (Horizontal Forehead Lines, Glabellar Frown Lines, and Lateral Canthal Lines)
Brief Title: Safety and Efficacy Study of the Simultaneous Treatment of Upper Facial Lines (Horizontal Forehead Lines, Glabellar Frown Lines and Crows Feet) in Subjects With Moderate to Severe Upper Facial Lines
Acronym: ULTRA II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Collaborators: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M602011070; 2019-004113-13 (EudraCT Number)
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-06

CONDITIONS: Moderate to Severe Upper Facial Lines (Horizontal Forehead Lines, Glabellar Frown Lines, and Lateral Canthal Lines)
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Main Period: Placebo (Group P) (Placebo Comparator): Subjects will receive placebo injection in all three UFL (GFL, HFL and LCL) on Day 1 of main period.
  Interventions: Drug: Placebo
- Main Period: NT 201 (Group U) (Experimental): Subjects will receive a total of 64 Units (U) of NT 201: 20 U of NT 201 injection both in the GFL area and in the HFL area, and 24 U of NT 201 injection in the LCL area (12 U per side) on Day 1 of main period.
  Interventions: Drug: NT 201
- Main Period: NT 201 and Placebo (Group L) (Experimental): Subjects will receive a total of 24 U NT 201: placebo injection both in the GFL and HFL area, and 24 U NT 201 injection in the LCL area (12 U per side) on Day 1 of main period.
  Interventions: Drug: NT 201; Drug: Placebo
- OLEX: NT 201 (Main Period: Group P) (Experimental): Subjects will receive a total of 64 U of NT 201: 20 U of NT 201 injection both in the GFL and in the HFL area, and 24 U of NT 201 injection in the LCL area (12 U per side) on Day 1 (Visit 8) and Visit 13 of OLEX period.
  Interventions: Drug: NT 201
- OLEX: NT 201 (Main Period: Group U) (Experimental): Subjects will receive a total of 64 U of NT 201: 20 U of NT 201 injection both in the GFL and in the HFL area, and 24 U of NT 201 injection in the LCL area (12 U per side) on Day 1 (Visit 8) and Visit 13 of OLEX period.
  Interventions: Drug: NT 201
- OLEX: NT 201 (Main Period: Group L) (Experimental): Subjects will receive a total of 64 U of NT 201: 20 U of NT 201 injection both in the GFL and in the HFL area, and 24 U of NT 201 injection in the LCL area (12 U per side) on Day 1 (Visit 8) and Visit 13 of OLEX period.
  Interventions: Drug: NT 201

INTERVENTIONS:
Drug: NT 201 — Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl).
  Other Names: IncobotulinumtoxinA; Xeomin; Botulinum toxin type A (150 kiloDalton), free from complexing protein
  Arms: Main Period: NT 201 (Group U); Main Period: NT 201 and Placebo (Group L); OLEX: NT 201 (Main Period: Group L); OLEX: NT 201 (Main Period: Group P); OLEX: NT 201 (Main Period: Group U)
Drug: Placebo — Solution for injection prepared by reconstitution of powder with percent (%) Sodium Chloride (NaCl).
  Arms: Main Period: NT 201 and Placebo (Group L); Main Period: Placebo (Group P)

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of NT 201 (active ingredient: Botulinum (neuro)toxin type A, free from complexing proteins) in the combined treatment of wrinkles in the upper face (Upper Facial Lines [UFL]): Horizontal Forehead Lines [HFL], Glabellar Frown Lines [GFL], and Lateral Canthal Lines [LCL]). It is a prospective, randomized, double-blind, placebo-controlled, multicenter study with a placebo-control main period (MP) followed by an open-label extension (OLEX) period.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients (male or female) 18 years of age or older.
* Horizontal forehead lines (HFL), glabellar frown lines (GFL), and symmetrical lateral canthal lines (LCL) of moderate to severe intensity at maximum contraction as assessed by the investigator and subject according to Merz Aesthetics Scales (MAS).

Exclusion Criteria:

* Previous treatment with botulinum neurotoxin (BoNT) of any serotype in the face within the last 12 months before injection.
* Any facial cosmetic procedure within the last 12 months before baseline injection.
* Previous treatment with any biodegradable filler in the face within the last 12 months before injection.
* Any previous insertion of permanent material in the face (regardless of the time between previous treatment and this study).
* Any medical condition that may put the subject at increased risk with exposure to NT201.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (10):
- Germany (10):
  - Merz Investigational Site, Bad Soden
  - Merz Investigational Site, Berlin
  - Merz Investigational Site, Bochum
  - Merz Investigational Site, Drensteinfurt
  - Merz Investigational Site, Düsseldorf
  - Merz Investigational Site, Hamburg
  - Merz Investigational Site, Mannheim
  - Merz Investigational Site, München
  - Merz Investigational Site, Potsdam
  - Merz Investigational Site, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pavicic T, Burgess C, Fabi S, Nestor MS, Bee EK, Imhof M, Dersch H, Sudimac V. Aesthetic Improvements Over Time: Long-Term Efficacy and Additional Outcomes of IncobotulinumtoxinA in the Simultaneous Treatment of Upper Facial Lines. J Cosmet Dermatol. 2025 Sep;24(9):e70460. doi: 10.1111/jocd.70460. PMID 40968493
- [Derived] Joseph J, Sudimac V, Mersmann S, Kerscher M. IncobotulinumtoxinA in the Treatment of Upper Facial Lines: Results From Two Randomized, Double-Blind, Placebo-Controlled, Phase III Studies. Aesthet Surg J. 2025 Feb 18;45(3):293-304. doi: 10.1093/asj/sjae222. PMID 39475143

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 12 investigational sites in Germany.
Pre-assignment Details: Of the 395 screened, 27 subjects exited as screen failures and 368 were randomized and enrolled to receive treatment with NT 201 or placebo in the main period of the study. Out of 358 subjects who completed the main period, 346 received treatment in the open-label extension (OLEX) period. As planned, participants (instead of facial lines) were assigned to the treatment groups and were assessed and analyzed. Therefore, data for participants is presented.
Groups:
- Main Period: Placebo (Group P): Subjects received placebo injection in all three upper facial lines (UFL) (glabellar frown lines [GFL], horizontal forehead lines [HFL] and lateral canthal lines [LCL]) on Day 1 of main period.
- Main Period: NT 201 (Group U): Subjects received a total of 64 Units (U) of NT 201: 20 U of NT 201 injection both in the GFL area and in the HFL area, and 24 U of NT 201 injection in the LCL area (12 U per side) on Day 1 of main period.
- Main Period: NT 201 and Placebo (Group L): Subjects received a total of 24 U NT 201: placebo injection both in the GFL and HFL area, and 24 U NT 201 injection in the LCL area (12 U per side) on Day 1 of main period.
- OLEX: NT 201 (Main Period: Group P); OLEX: NT 201 (Main Period: Group U); OLEX: NT 201 (Main Period: Group L): Subjects received a total of 64 U of NT 201: 20 U of NT 201 injection both in the GFL and in the HFL area, and 24 U of NT 201 injection in the LCL area (12 U per side) on Day 1 (Visit 8) and Visit 13 of OLEX period.
Period: Main Period (Up to 22 Weeks)
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U) | Main Period: NT 201 and Placebo (Group L) | OLEX: NT 201 (Main Period: Group P) | OLEX: NT 201 (Main Period: Group U) | OLEX: NT 201 (Main Period: Group L)
Started | 94 | 184 | 90 | 0 | 0 | 0
Completed | 91 | 180 | 87 | 0 | 0 | 0
Not Completed | 3 | 4 | 3 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0 | 0 | 0
Period: OLEX Period (Up to 39 Weeks)
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U) | Main Period: NT 201 and Placebo (Group L) | OLEX: NT 201 (Main Period: Group P) | OLEX: NT 201 (Main Period: Group U) | OLEX: NT 201 (Main Period: Group L)
Started | 0 | 0 | 0 | 89 (Several subjects who completed main period did not receive treatment in the OLEX period due to non-eligibility or other reasons.) | 170 (Several subjects who completed main period did not receive treatment in the OLEX period due to non-eligibility or other reasons.) | 87 (Several subjects who completed main period did not receive treatment in the OLEX period due to non-eligibility or other reasons.)
Completed | 0 | 0 | 0 | 81 | 156 | 76
Not Completed | 0 | 0 | 0 | 8 | 14 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 3 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other eligibility criteria for re-injection not met | 0 | 0 | 0 | 1 | 0 | 0
Not completed — No need for re-injection | 0 | 0 | 0 | 1 | 9 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 5 | 4
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized subjects.
Groups:
- Main Period: Placebo (Group P): Subjects received placebo injection in all three UFL (GFL, HFL and LCL) on Day 1 of main period.
- Main Period: NT 201 (Group U): Subjects received a total of 64 U of NT 201: 20 U of NT 201 injection both in the GFL area and in the HFL area, and 24 U of NT 201 injection in the LCL area (12 U per side) on Day 1 of main period.
- Total: Total of all reporting groups
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U) | Main Period: NT 201 and Placebo (Group L) | Total
Number analyzed (Participants) | 94 | 184 | 90 | 368
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (9.15) | 46.0 (9.92) | 45.9 (9.88) | 45.7 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 147 | 72 | 303
  Male | 10 | 37 | 18 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 93 | 182 | 88 | 363
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 94 | 182 | 89 | 365
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Main Period: Percentage of Glabellar Frown Line (GFL) Responders at Day 30
Description: The Merz aesthetics scales (MAS) are 5-point scales used to identify responders in a clinical context. They are validated photograph-based outcome instruments designed specifically for assessment of each upper facial area. GFL-response was defined as a score of 0 (no) or 1 (mild) and at least two-grade improvement from baseline to Day 30 of main period on MAS for GFL at maximum contraction as assessed by both the investigator and the subject. The MAS for GFL ranged as 0 to 4 where 0 is "No glabellar lines", 1 is "Mild glabellar lines", 2 is "Moderate glabellar lines", 3 is "Severe glabellar lines" and 4 is "Very severe glabellar lines".
Time Frame: Day 30
Population: Target population of main primary estimand included subjects with HFL, GFL and LCL of moderate to severe intensity at maximum contraction as assessed by investigator and subject according to MAS, as randomized in this study: Subset of subjects randomized to UFL (Group U) or to placebo (Group P) groups, grouped by randomized treatment assignment.
Measure: Number; unit: percentage of subjects
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U)
Number analyzed (Participants) | 94 | 182
percentage of subjects | 0 | 49.5
Statistical Analysis 1: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 (Group U); Test type: Superiority; p < 0.0001, Mantel Haenszel

2. Primary Outcome: Main Period: Percentage of Horizontal Forehead Lines (HFL) Responders at Day 30
Description: The MAS are 5-point scales used to identify responders in a clinical context. They are validated photograph-based outcome instruments designed specifically for assessment of each upper facial area. HFL-response was defined as a score of 0 (no) or 1 (mild) and at least two-grade improvement from baseline to Day 30 of main period on MAS for HFL at maximum contraction as assessed by both the investigator and the subject. The MAS for HFL ranged as 0 to 4 where 0 is "No lines", 1 is "Mild lines", 2 is "Moderate lines", 3 is "Severe lines" and 4 is "Very severe lines".
Time Frame: Day 30
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U)
Number analyzed (Participants) | 94 | 182
percentage of subjects | 0 | 57.7
Statistical Analysis 1: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 (Group U); Test type: Superiority; p < 0.0001, Mantel Haenszel

3. Primary Outcome: Main Period: Percentage of Lateral Canthal Lines (LCL) Responders at Day 30
Description: The MAS are 5-point scales used to identify responders in a clinical context. They are validated photograph-based outcome instruments designed specifically for assessment of each upper facial area. LCL-response was defined as a score of 0 (no) or 1 (mild) and at least two-grade improvement from baseline to Day 30 of main period on MAS for both left and right LCL at maximum contraction as assessed by both the investigator and the subject. The MAS for LCL ranged as 0 to 4 where 0 is "No lines", 1 is "Mild lines", 2 is "Moderate lines", 3 is "Severe lines" and 4 is "Very severe lines".
Time Frame: Day 30
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U)
Number analyzed (Participants) | 94 | 182
percentage of subjects | 0 | 32.4
Statistical Analysis 1: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 (Group U); Test type: Superiority; p < 0.0001, Mantel Haenszel

4. Secondary Outcome: Main Period: Percentage of Subjects With a Score of 0 (no) or 1 (Mild) on MAS for GFL at Maximum Contraction as Assessed by the Investigator at Day 30
Description: The MAS are 5-point scales used to identify responders in clinical context. They are validated photograph-based outcome instruments designed specifically for assessment of each upper facial area. MAS for GFL ranged as 0 to 4, where 0 is "No glabellar lines", 1 is "Mild glabellar lines", 2 is "Moderate glabellar lines", 3 is "Severe glabellar lines" and 4 is "Very severe glabellar lines".
Time Frame: Day 30
Population: Target population of main key secondary estimand included subjects with HFL, GFL and LCL of moderate to severe intensity at maximum contraction as assessed by investigator and subject according to MAS, as randomized in this study: Subset of subjects randomized to UFL (Group U) or to placebo (Group P) groups, grouped by randomized treatment assignment.
Measure: Number; unit: percentage of subjects
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U)
Number analyzed (Participants) | 94 | 182
percentage of subjects | 0.0 | 86.8
Statistical Analysis 1: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 (Group U); Test type: Superiority; p < 0.0001, Mantel Haenszel

5. Secondary Outcome: Main Period: Percentage of Subjects With a Score of 0 (no) or 1 (Mild) on MAS for HFL at Maximum Contraction as Assessed by the Investigator at Day 30
Description: The MAS are 5-point scales used to identify responders in clinical context. They are validated photograph-based outcome instruments designed specifically for assessment of each upper facial area. The MAS for HFL ranged as 0 to 4 where 0 is "No lines", 1 is "Mild lines", 2 is "Moderate lines", 3 is "Severe lines" and 4 is "Very severe lines".
Time Frame: Day 30
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U)
Number analyzed (Participants) | 94 | 182
percentage of subjects | 1.1 | 86.3
Statistical Analysis 1: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 (Group U); Test type: Superiority; p < 0.0001, Mantel Haenszel

6. Secondary Outcome: Main Period: Percentage of Subjects With a Score of 0 (no) or 1 (Mild) on MAS for Both Left and Right LCL at Maximum Contraction as Assessed by the Investigator at Day 30
Description: The MAS are 5-point scales used to identify responders in clinical context. They are validated photograph-based outcome instruments designed specifically for assessment of each upper facial area. The MAS for LCL ranged as 0 to 4 where 0 is "No lines", 1 is "Mild lines", 2 is "Moderate lines", 3 is "Severe lines" and 4 is "Very severe lines".
Time Frame: Day 30
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U)
Number analyzed (Participants) | 94 | 182
percentage of subjects | 2.1 | 75.8
Statistical Analysis 1: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 (Group U); Test type: Superiority; p < 0.0001, Mantel Haenszel

7. Secondary Outcome: Main Period: Percentage of Subjects With a Score of 0 (no) or 1 (Mild) on MAS for GFL at Maximum Contraction as Assessed by the Subject at Day 30
Description: The MAS are 5-point scales used to identify responders in clinical context. They are validated photograph-based outcome instruments designed specifically for assessment of each upper facial area. The MAS for GFL ranged as 0 to 4, where 0 is "No glabellar lines", 1 is "Mild glabellar lines", 2 is "Moderate glabellar lines", 3 is "Severe glabellar lines" and 4 is "Very severe glabellar lines".
Time Frame: Day 30
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U)
Number analyzed (Participants) | 94 | 182
percentage of subjects | 1.1 | 73.6
Statistical Analysis 1: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 (Group U); Test type: Superiority; p < 0.0001, Mantel Haenszel

8. Secondary Outcome: Main Period: Percentage of Subjects With a Score of 0 (no) or 1 (Mild) on MAS for HFL at Maximum Contraction as Assessed by the Subject at Day 30
Description: as for outcome 5
Time Frame: Day 30
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U)
Number analyzed (Participants) | 94 | 182
percentage of subjects | 2.1 | 79.1
Statistical Analysis 1: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 (Group U); Test type: Superiority; p < 0.0001, Mantel Haenszel

9. Secondary Outcome: Main Period: Percentage of Subjects With a Score of 0 (no) or 1 (Mild) on MAS for Both Left and Right LCL at Maximum Contraction as Assessed by the Subject at Day 30
Description: as for outcome 6
Time Frame: Day 30
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U)
Number analyzed (Participants) | 94 | 182
percentage of subjects | 3.2 | 65.4
Statistical Analysis 1: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 (Group U); Test type: Superiority; p < 0.0001, Mantel Haenszel

10. Secondary Outcome: Main Period: Global Aesthetic Improvement Scale (GAIS) at Day 30 as Assessed by the Subjects
Description: The GAIS is a 7-point Likert scale capturing the global aesthetic improvement ranging from +3 (very much improved); +2 (much improved); +1 (improved); 0 (no change); -1 (worse); -2 (much worse); -3 (very much worse), as assessed by the subject. GAIS as assessed by the subject at Day 30 was analyzed using an analysis of covariance (ANCOVA) model.
Time Frame: Day 30
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U)
Number analyzed (Participants) | 94 | 182
score on a scale | 0.02 [-0.11 to 0.15] | 2.00 [1.90 to 2.09]
Statistical Analysis 1: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 (Group U); Test type: Superiority; p < 0.0001, ANCOVA

11. Secondary Outcome: Main Period: Percentage of Subjects With at Least One-grade Improvement From Baseline to Day 30 of Main Period on MAS for GFL at Maximum Contraction as Assessed by the Investigator
Description: The MAS are 5-point scales used to identify responders in a clinical context. They are validated photograph- based outcome instruments designed specifically for assessment of each upper facial area. The MAS for GFL ranged as 0 to 4 where 0 is "No glabellar lines", 1 is "Mild glabellar lines", 2 is "Moderate glabellar lines", 3 is "Severe glabellar lines" and 4 is "Very severe glabellar lines".
Time Frame: Day 30
Population: FAS. Here "overall number of subjects analyzed" were subjects who had non-missing data for this outcome measure.
Measure: Number; unit: percentage of subjects
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U) | Main Period: NT 201 and Placebo (Group L)
Number analyzed (Participants) | 91 | 181 | 88
percentage of subjects | 5.5 | 96.7 | 4.5
Statistical Analysis 1: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 (Group U); Test type: Superiority; p < 0.0001, Mantel Haenszel

12. Secondary Outcome: Main Period: Percentage of Subjects With at Least One-grade Improvement From Baseline to Day 30 of Main Period on MAS for HFL at Maximum Contraction as Assessed by the Investigator
Description: The MAS are 5-point scales used to identify responders in a clinical context. They are validated photograph-based outcome instruments designed specifically for assessment of each upper facial area. The MAS for HFL ranged as 0 to 4 where 0 is "No lines", 1 is "Mild lines", 2 is "Moderate lines", 3 is "Severe lines" and 4 is "Very severe lines".
Time Frame: Day 30
Population: FAS. Here "overall number of subjects analyzed" were subjects who had non-missing data for this outcome measure.
Measure: Number; unit: percentage of subjects
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U) | Main Period: NT 201 and Placebo (Group L)
Number analyzed (Participants) | 91 | 181 | 88
percentage of subjects | 3.3 | 96.1 | 3.4
Statistical Analysis 1: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 (Group U); Test type: Superiority; p < 0.0001, Mantel Haenszel

13. Secondary Outcome: Main Period: Percentage of Subjects With at Least One-grade Improvement From Baseline to Day 30 of Main Period on MAS for Both Left and Right LCL at Maximum Contraction as Assessed by the Investigator
Description: The MAS are 5-point scales used to identify responders in a clinical context. They are validated photograph-based outcome instruments designed specifically for assessment of each upper facial area. The MAS for LCL ranged as 0 to 4 where 0 is "No lines", 1 is "Mild lines", 2 is "Moderate lines", 3 is "Severe lines" and 4 is "Very severe lines".
Time Frame: Day 30
Population: FAS. Here "overall number of subjects analyzed" were subjects who had non-missing data for this outcome measure.
Measure: Number; unit: percentage of subjects
Groups:
- Main Period: NT 201 and Placebo (Group L): Subjects received placebo a total of 24 U NT 201: injection both in the GFL and HFL area, and 24 U NT 201 injection in the LCL area (12 U per side) on Day 1 of main period.
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U) | Main Period: NT 201 and Placebo (Group L)
Number analyzed (Participants) | 91 | 181 | 88
percentage of subjects | 8.8 | 91.7 | 68.2
Statistical Analysis 1: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 (Group U); Test type: Superiority; p < 0.0001, Mantel Haenszel
Statistical Analysis 2: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 and Placebo (Group L); Test type: Superiority; p < 0.0001, Mantel Haenszel

14. Secondary Outcome: Main Period: Global Aesthetic Improvement Scale (GAIS) at Day 30 as Assessed by the Investigator
Description: The GAIS is a 7-point Likert scale capturing the global aesthetic improvement ranging from +3 (very much improved); +2 (much improved); +1 (improved); 0 (no change); -1 (worse); -2 (much worse); -3 (very much worse), as assessed by the investigator. GAIS as assessed by the investigator at Day 30 was analyzed using an ANCOVA model.
Time Frame: Day 30
Population: FAS. Here "overall number of subjects analyzed" were subjects who had non-missing data for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U) | Main Period: NT 201 and Placebo (Group L)
Number analyzed (Participants) | 91 | 181 | 88
score on a scale | 0.03 [-0.09 to 0.14] | 2.23 [2.14 to 2.31] | 0.68 [0.56 to 0.80]
Statistical Analysis 1: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 (Group U); Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Main Period: Placebo (Group P) vs Main Period: NT 201 and Placebo (Group L); Test type: Superiority; p < 0.0001, ANCOVA

15. Secondary Outcome: Main Period: Number of Subjects With Related Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs during the Main Period are defined as adverse events (AEs) with onset or worsening on or after date and time of first dose of study treatment and before date and time of first administration of study treatment in the OLEX period or the final study visit, if subject was not treated in the OLEX period. An AE is considered to be related if a causal relationship between study treatment and the AE is at least reasonably possible.
Time Frame: Up to 22 weeks
Population: The Safety Evaluation Set (SES) included all subjects treated.
Measure: Count of Participants; unit: Participants
Groups:
- Main Period: NT 201 (Group L): Subjects received a total of 24 U NT 201: placebo injection both in the GFL and HFL area, and 24 U NT 201 injection in the LCL area (12 U per side) on Day 1 of main period.
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U) | Main Period: NT 201 (Group L)
Number analyzed (Participants) | 94 | 184 | 90
Participants | 12 | 35 | 10

16. Secondary Outcome: OLEX: Number of Subjects With Related TEAEs
Description: TEAEs of the OLEX period are defined as adverse events (AEs) with onset or worsening on or after date and time of first dose of study treatment in the OLEX period up to and including the final study visit. An AE is considered to be related if a causal relationship between study treatment and the AE is at least reasonably possible.
Time Frame: Up to 39 weeks
Population: SES.
Measure: Count of Participants; unit: Participants
Arm/Group | OLEX: NT 201 (Main Period: Group P) | OLEX: NT 201 (Main Period: Group U) | OLEX: NT 201 (Main Period: Group L)
Number analyzed (Participants) | 89 | 170 | 87
Participants | 18 | 32 | 12

ADVERSE EVENTS:
Time Frame: Main Period: Up to 22 weeks; OLEX Period: Up to 39 weeks
Description: SES. The investigator reported AEs systematically at each visit.
Arm/Group | Main Period: Placebo (Group P) | Main Period: NT 201 (Group U) | Main Period: NT 201 and Placebo (Group L) | OLEX: NT 201 (Main Period: Group P) | OLEX: NT 201 (Main Period: Group U) | OLEX: NT 201 (Main Period: Group L)
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/184 | 0/90 | 0/89 | 0/170 | 0/87
Serious Adverse Events (participants affected / at risk) | 4/94 | 1/184 | 2/90 | 2/89 | 6/170 | 3/87
Other Adverse Events (participants affected / at risk) | 23/94 | 43/184 | 23/90 | 39/89 | 74/170 | 29/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Period: Placebo (Group P) (N=94) | Main Period: NT 201 (Group U) (N=184) | Main Period: NT 201 and Placebo (Group L) (N=90) | OLEX: NT 201 (Main Period: Group P) (N=89) | OLEX: NT 201 (Main Period: Group U) (N=170) | OLEX: NT 201 (Main Period: Group L) (N=87)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1 | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Post-acute COVID-19 syndrome (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intracranial hypotension (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Period: Placebo (Group P) (N=94) | Main Period: NT 201 (Group U) (N=184) | Main Period: NT 201 and Placebo (Group L) (N=90) | OLEX: NT 201 (Main Period: Group P) (N=89) | OLEX: NT 201 (Main Period: Group U) (N=170) | OLEX: NT 201 (Main Period: Group L) (N=87)
Nasopharyngitis (Infections and infestations) | 4 | 3 | 3 | 9 | 22 | 11
COVID-19 (Infections and infestations) | 4 | 2 | 0 | 13 | 33 | 12
Injection site haematoma (General disorders) | 8 | 15 | 9 | 11 | 22 | 9
Headache (Nervous system disorders) | 8 | 18 | 7 | 9 | 9 | 2
Immunisation reaction (Immune system disorders) | 2 | 10 | 9 | 4 | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT04622254/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT04622254/SAP_001.pdf